CLINICAL TRIAL: NCT03179345
Title: A Phase 4, Double-Blind, Placebo-Controlled, Crossover Study Comparing Simulated Driving Performance, Daytime Sedation, and Cognition in Healthy Volunteers Taking Therapeutic Doses of Gralise®, Neurontin®, or Lyrica®
Brief Title: Simulated Driving Performance, Daytime Sedation and Cognition in Healthy Volunteers Taking Gralise, Neurontin or Lyrica
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Other
Other Study IDs: GRAL-PX-8401
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: Volunteer; Pharmacodynamics; Pharmacokinetics
MeSH Terms: interventions — Gabapentin; Pregabalin; Sugars

ARMS (4):
- Gralise® (gabapentin) (Active Comparator): Gralise® 3 x 600 mg tablets (1800 mg total dose) administered once daily at 7:00 pm on Day 1 and Day 2 with one placebo capsule matching the over-encapsulation of doses of Neurontin® and Lyrica®. At other dosing times, treatment consisted of 3 placebo tablets matching the appearance of Gralise® and 1 placebo capsule.
  Interventions: Drug: Gabapentin
- Neurontin® (gabapentin) (Active Comparator): Neurontin® 1 x 600 mg film-coated tablet administered 3 times daily at 7:00 pm on Day 1, at 8:00 am, 2:00 pm and 8:00 pm on Day 2 and at 8:00 a.m. on Day 3. Each dose of Neurontin® was over-encapsulated and administered with 3 placebo tablets matching the appearance of Gralise®.
  Interventions: Drug: Gabapentin
- Lyrica® (pregabalin) (Active Comparator): Lyrica® 1 x 150 mg capsule administered 2 times daily at 7:00 pm on Day 1, at 8:00 am and 8:00 pm on Day 2 and at 8:00 a.m. on Day 3. Each dose of Lyrica® was over-encapsulated and administered with 3 placebo tablets matching the appearance of Gralise®.
  Interventions: Drug: Pregabalin
- Placebo (sugar pill) (Placebo Comparator): Each dose consisted of 3 placebo tablets matching the appearance of Gralise® and 1 placebo capsule matching the over-encapsulation of doses of Neurontin® and Lyrica®.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gabapentin
  Other Names: Gralise®, Neurontin®
  Arms: Gralise® (gabapentin); Neurontin® (gabapentin)
Drug: Pregabalin
  Other Names: Lyrica®
  Arms: Lyrica® (pregabalin)
Other: Placebo
  Other Names: Sugar Pill
  Arms: Placebo (sugar pill)

SUMMARY:
Phase 4, double-blind, placebo-controlled, four treatment, four sequence crossover study comparing simulated driving performance, daytime sedation and cognition in healthy volunteers administered therapeutic doses of Gralise® (Treatment A), Neurontin® (Treatment B), Lyrica® (Treatment C) and placebo (Treatment D). All doses were administered under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Between 40 and 80 years of age, inclusive.
* Body weight > 50 kg and BMI between 18 and 32 kg/m2, inclusive.
* Able to give informed consent.
* Licensed, experienced driver who had driven at least 3 times a week for the past 3 years and had visual acuity adequate for driving, as assessed by the investigator or designee.
* Able to complete a 1 hour simulated driving test and demonstrate satisfactory driving skills, as determined by the investigator or designee.
* Karolinska Sleep Scale (KSS) score of <=5.
* Other criteria apply.

Exclusion Criteria:

* Known history of allergic reaction, hypersensitivity or clinically significant intolerance to gabapentin, pregabalin or any pharmaceutical materials, or any of the ingredients in the protocol-specified meals.
* Pregnant or lactating or considered at risk of pregnancy.
* Any medical condition or any laboratory abnormality or ECG abnormality that would, in the opinion of the investigator, contraindicate study participation.
* Impaired liver function (e.g., alanine aminotransferase [ALT] ≥2 times the upper limit of normal [ULN] or bilirubin ≥2 times ULN), known active hepatic disease (e.g., hepatitis), or evidence of clinically significant liver disease or other condition affecting the liver that may suggest the potential for an increased susceptibility to hepatic toxicity with oral gabapentin or pregabalin exposure.
* Any history of renal disease that, in the opinion of the investigator, would contraindicate study participation; or subject had significantly impaired renal function as evidenced by an estimated GFR of ≤ 80 ml/min/1.73m2.
* History or evidence of a sleep disorder, including sleep apnea (obstructive, central or mixed), narcolepsy or primary insomnia.
* Other criteria apply.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2015-11-20 (Actual); Study Completion 2015-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of R&D, Study Director — Depomed

REFERENCES:
- [Derived] Schmidt P, Rao S. Effects of gabapentin, pregabalin and gastroretentive gabapentin on simulated driving, daytime sedation and cognition. Pain Manag. 2018 Jul 1;8(4):297-306. doi: 10.2217/pmt-2018-0005. Epub 2018 Apr 19. PMID 29671676

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 32 healthy subjects enrolled in this crossover study. Each subject was randomly assigned to 1 out of 4 treatment sequences.
  Abbreviations:
  Gral = Gralise®; Neur = Neurontin®; Lyr = Lyrica®; Plbo = Placebo.
Groups:
- Gral First, Then Neur, Lyr, and Plbo: Gralise® (gabapentin) 3 x 600 mg tablets (1800 mg total): Dosed once daily in the evening on Day 1 and Day 2.
  Neurontin® (gabapentin) 1 x 600 mg film-coated tablet: Dosed 3 times daily starting in the evening on Day 1, in the morning, afternoon, and evening on Day 2, and in the morning on Day 3.
  Lyrica® (pregabalin) 1 x 150 mg capsule: Dosed 2 times daily starting in the evening on Day 1, in the morning and evening on Day 2, and in the morning on Day 3.
  Placebo (sugar pill): Three (3) placebo tablets matching the appearance of Gralise® & 1 placebo capsule matching the over-encapsulation of doses of Neurontin® & Lyrica®.
  All treatments were administered following a meal.
  Each treatment period was separated by a 7-day washout interval.
- Neur First, Then Plbo, Gral, and Lyr: Neurontin® (gabapentin) 1 x 600 mg film-coated tablet: Dosed 3 times daily starting in the evening on Day 1, in the morning, afternoon, and evening on Day 2, and in the morning on Day 3.
  Placebo (sugar pill): Three (3) placebo tablets matching the appearance of Gralise® & 1 placebo capsule matching the over-encapsulation of doses of Neurontin® & Lyrica®.
  Gralise® (gabapentin) 3 x 600 mg tablets (1800 mg total): Dosed once daily in the evening on Day 1 and Day 2.
  Lyrica® (pregabalin) 1 x 150 mg capsule: Dosed 2 times daily starting in the evening on Day 1, in the morning and evening on Day 2, and in the morning on Day 3.
  All treatments were administered following a meal.
  Each treatment period was separated by a 7-day washout interval.
- Lyr First, Then Gral, Plbo, and Neur: Lyrica® (pregabalin) 1 x 150 mg capsule: Dosed 2 times daily starting in the evening on Day 1, in the morning and evening on Day 2, and in the morning on Day 3.
  Gralise® (gabapentin) 3 x 600 mg tablets (1800 mg total): Dosed once daily in the evening on Day 1 and Day 2.
  Placebo (sugar pill): Three (3) placebo tablets matching the appearance of Gralise® & 1 placebo capsule matching the over-encapsulation of doses of Neurontin® & Lyrica®.
  Neurontin® (gabapentin) 1 x 600 mg film-coated tablet: Dosed 3 times daily starting in the evening on Day 1, in the morning, afternoon, and evening on Day 2, and in the morning on Day 3.
  All treatments were administered following a meal.
  Each treatment period was separated by a 7-day washout interval.
- Plbo First, Then Lyr, Neur, and Gral: Placebo (sugar pill): Three (3) placebo tablets matching the appearance of Gralise® & 1 placebo capsule matching the over-encapsulation of doses of Neurontin® & Lyrica®.
  Lyrica® (pregabalin) 1 x 150 mg capsule: Dosed 2 times daily starting in the evening on Day 1, in the morning and evening on Day 2, and in the morning on Day 3.
  Neurontin® (gabapentin) 1 x 600 mg film-coated tablet: Dosed 3 times daily starting in the evening on Day 1, in the morning, afternoon, and evening on Day 2, and in the morning on Day 3.
  Gralise® (gabapentin) 3 x 600 mg tablets (1800 mg total): Dosed once daily in the evening on Day 1 and Day 2.
  All treatments were administered following a meal.
  Each treatment period was separated by a 7-day washout interval.
Period: Overall Study
Arm/Group | Gral First, Then Neur, Lyr, and Plbo | Neur First, Then Plbo, Gral, and Lyr | Lyr First, Then Gral, Plbo, and Neur | Plbo First, Then Lyr, Neur, and Gral
Started | 8 | 8 | 8 | 8
Received Gralise® | 8 | 7 | 7 | 6
Received Neurontin® | 8 | 8 | 7 | 8
Received Lyrica® | 8 | 7 | 8 | 8
Received Placebo | 8 | 7 | 7 | 8
Completed | 8 | 7 | 7 | 6
Not Completed | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gral First, Then Neur, Lyr, and Plbo | Neur First, Then Plbo, Gral, and Lyr | Lyr First, Then Gral, Plbo, and Neur | Plbo First, Then Lyr, Neur, and Gral | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (5.32) | 47.6 (5.29) | 51.0 (9.35) | 46.8 (4.06) | 48.6 (6.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 1 | 8
  Male | 7 | 5 | 5 | 7 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the "Standard Deviation of the Lateral Position" (SDLP) Measured on the Driving Simulator Between Gralise® and Neurontin®
Description: SDLP (feet): This is a measurement of change from maintaining the normal driving position in the lane over time and / or distance.
Time Frame: Baseline and Hour 3 on Day 3
Population: The above is the only Primary Outcome Measure (comparing the SDLP between Gralise® and Neurontin®).
Measure: Least Squares Mean (Standard Error); unit: feet
Groups:
- Gralise® (Gabapentin): Gralise® (gabapentin) 3 x 600 mg tablets (1800 mg total): Dosed once daily in the evening on Day 1 and Day 2.
- Neurontin® (Gabapentin): Neurontin® (gabapentin) 1 x 600 mg film-coated tablet: Dosed 3 times daily starting in the evening on Day 1, in the morning, afternoon, and evening on Day 2, and in the morning on Day 3.
- Placebo: Each dose consisted of 3 placebo tablets matching the appearance of Gralise® and 1 placebo capsule matching the over-encapsulation of doses of Neurontin® and Lyrica®: Dosed 3 times daily starting in the evening on Day 1, in the morning, afternoon, and evening on Day 2, and in the morning on Day 3.
Arm/Group | Gralise® (Gabapentin) | Neurontin® (Gabapentin) | Placebo
Number analyzed (Participants) | 28 | 31 | 30
feet | 0.255 (0.0781) | 0.395 (0.0763) | 0.135 (0.0770)
Statistical Analysis 1: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Test type: Superiority; p = 0.0275, ANOVA; Mixed model including terms for sequence, study treatment, and period as fixed effects and subject nested within Sequence as a random effect; Mean Difference (Net) = -0.141, 95% CI 2-sided [-0.266 to -0.016], Standard Error of Mean 0.06 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 2: Comparison: Gralise® (Gabapentin) vs Placebo; Test type: Superiority; p = 0.0611, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.120, 95% CI 2-sided [-0.006 to 0.245], Standard Error of Mean 0.06 — SE of difference estimated by dividing width of 95% CI by 4

2. Secondary Outcome: Change From Baseline in the "Standard Deviation of the Lateral Position" (SDLP) Measured on the Driving Simulator Between Gralise® and Lyrica®
Description: as for outcome 1
Time Frame: Baseline and Hour 3 on Day 3
Population: The above is a Secondary Outcome Measure (comparing the SDLP between Gralise® and Lyrica®).
Measure: Least Squares Mean (Standard Error); unit: feet
Groups:
- Lyrica® (Pregabalin): Lyrica® (pregabalin) 1 x 150 mg capsule: Dosed 2 times daily starting in the evening on Day 1, in the morning and evening on Day 2, and in the morning on Day 3.
Arm/Group | Gralise® (Gabapentin) | Lyrica® (Pregabalin) | Placebo
Number analyzed (Participants) | 28 | 30 | 30
feet | 0.255 (0.0781) | 0.356 (0.0770) | 0.135 (0.0770)
Statistical Analysis 1: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Test type: Superiority; p = 0.1103, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.102, 95% CI 2-sided [-0.227 to 0.024], Standard Error of Mean 0.06 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 2: Comparison: Gralise® (Gabapentin) vs Placebo; Test type: Superiority; p = 0.0611, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.120, 95% CI 2-sided [-0.006 to 0.245], Standard Error of Mean 0.06 — SE of difference estimated by dividing width of 95% CI by 4

3. Secondary Outcome: Change From Baseline Between, Gralise® and Neurontin®, Gralise® and Lyrica® for Cognitive Evaluation of Cogstate - Detection Task (DET)
Description: Cogstate - Detection Task (DET) is a simple reaction time test of Psychomotor Function. Higher change from baseline means better performance.
Time Frame: Baseline and Hour 3 on Day 3
Measure: Least Squares Mean (Standard Error); unit: msec
Groups:
- Gralise® (Gabapentin): Gralise® 3 x 600 mg tablets (1800 mg total dose) administered once daily at 7:00 pm on Day 1 and Day 2 with one placebo capsule matching the over-encapsulation of doses of Neurontin® and Lyrica®. At other dosing times, treatment consisted of 3 placebo tablets matching the appearance of Gralise® and 1 placebo capsule.
  Gabapentin
- Neurontin® (Gabapentin): Neurontin® 1 x 600 mg film-coated tablet administered 3 times daily at 7:00 pm on Day 1, at 8:00 am, 2:00 pm and 8:00 pm on Day 2 and at 8:00 a.m. on Day 3. Each dose of Neurontin® was over-encapsulated and administered with 3 placebo tablets matching the appearance of Gralise®.
  Gabapentin
- Lyrica® (Pregabalin): Lyrica® 1 x 150 mg capsule administered 2 times daily at 7:00 pm on Day 1, at 8:00 am and 8:00 pm on Day 2 and at 8:00 a.m. on Day 3. Each dose of Lyrica® was over-encapsulated and administered with 3 placebo tablets matching the appearance of Gralise®.
  Pregabalin
- Placebo (Sugar Pill): Each dose consisted of 3 placebo tablets matching the appearance of Gralise® and 1 placebo capsule matching the over-encapsulation of doses of Neurontin® and Lyrica®.
  Placebo
Arm/Group | Gralise® (Gabapentin) | Neurontin® (Gabapentin) | Lyrica® (Pregabalin) | Placebo (Sugar Pill)
Number analyzed (Participants) | 28 | 31 | 30 | 30
msec | 0.00 (0.013) | 0.00 (0.012) | -0.01 (0.012) | -0.00 (0.012)
Statistical Analysis 1: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Test type: Superiority; p = 0.9946, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.02 to 0.02], Standard Error of Mean 0.01 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 2: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Test type: Superiority; p = 0.1673, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.01 to 0.04], Standard Error of Mean 0.0125 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 3: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Test type: Superiority; p = 0.6208, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.02 to 0.03], Standard Error of Mean 0.0125 — SE of difference estimated by dividing width of 95% CI by 4

4. Secondary Outcome: Change From Baseline Between, Gralise® and Neurontin®, Gralise® and Lyrica® for Cognitive Evaluation of Cogstate - Groton Maze Learning Test (GMLT).
Description: Cogstate - The Groton Maze Learning test is a measure Executive Function. Total number of errors made while attempting to learn the same hidden pathway across the consecutive learning trials performed at a single assessment. Lower score means better performance. Higher change from baseline means better performance.
Time Frame: Baseline and Hour 3 on Day 3
Measure: Least Squares Mean (Standard Error); unit: Number of errors on test
Arm/Group | Gralise® (Gabapentin) | Neurontin® (Gabapentin) | Lyrica® (Pregabalin) | Placebo (Sugar Pill)
Number analyzed (Participants) | 28 | 31 | 30 | 30
Number of errors on test | -0.40 (2.484) | -0.01 (2.385) | -0.64 (2.419) | 3.32 (2.420)
Statistical Analysis 1: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Test type: Superiority; p = 0.8799, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.40, 95% CI 2-sided [-5.59 to 4.80], Standard Error of Mean 2.60 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 2: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Test type: Superiority; p = 0.9277, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.24, 95% CI 2-sided [-4.97 to 5.45], Standard Error of Mean 2.61 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 3: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Test type: Superiority; p = 0.1587, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -3.73, 95% CI 2-sided [-8.94 to 1.49] — SE of difference estimated by dividing width of 95% CI by 4

5. Secondary Outcome: Change From Baseline Between, Gralise® and Neurontin®, Gralise® and Lyrica® for Cognitive Evaluation of Cogstate - Identification Task (IDN).
Description: Cogstate - Identification Task (IDN) assesses Attention. Score is speed of performance (mean of the log10 transformed reaction times for correct responses). Lower score (quicker speed) is better performance. Higher change from baseline means better performance.
Time Frame: Baseline and Hour 3 on Day 3
Measure: Least Squares Mean (Standard Error); unit: Score on Scale
Arm/Group | Gralise® (Gabapentin) | Neurontin® (Gabapentin) | Lyrica® (Pregabalin) | Placebo (Sugar Pill)
Number analyzed (Participants) | 28 | 31 | 30 | 30
Score on Scale | -0.00 (0.000) | 0.00 (0.000) | -0.00 (0.000) | 0.01 (0.000)
Statistical Analysis 1: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Test type: Superiority; p = 0.7111, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.03 to 0.02], Standard Error of Mean 0.0125 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 2: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Test type: Superiority; p = 0.9048, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.02 to 0.02], Standard Error of Mean 0.01 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 3: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Test type: Superiority; p = 0.3262, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.03 to 0.01], Standard Error of Mean 0.01 — SE of difference estimated by dividing width of 95% CI by 4

6. Secondary Outcome: Change From Baseline Between, Gralise® and Neurontin®, Gralise® and Lyrica® for Cognitive Evaluation of Cogstate - International Shopping List Test (ISL)
Description: Cogstate - International Shopping List (ISL) test is a measure of verbal learning and uses a well-validated list-learning paradigm. Total number of correct responses remembering the word list on three consecutive trials at a single assessment. Higher score is better performance. Higher change from baseline means better performance.
Time Frame: Baseline and Hour 3 on Day 3
Measure: Least Squares Mean (Standard Error); unit: Score on Scale
Arm/Group | Gralise® (Gabapentin) | Neurontin® (Gabapentin) | Lyrica® (Pregabalin) | Placebo (Sugar Pill)
Number analyzed (Participants) | 28 | 31 | 30 | 30
Score on Scale | 0.36 (0.684) | 0.82 (0.648) | 0.03 (0.660) | -0.01 (0.660)
Statistical Analysis 1: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Test type: Superiority; p = 0.5950, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.46, 95% CI 2-sided [-2.18 to 1.26], Standard Error of Mean 0.860 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 2: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Test type: Superiority; p = 0.7057, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.33, 95% CI 2-sided [-1.40 to 2.06], Standard Error of Mean 0.865 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 3: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Test type: Superiority; p = 0.6741, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.37, 95% CI 2-sided [-1.36 to 2.10], Standard Error of Mean 0.865 — SE of difference estimated by dividing width of 95% CI by 4

7. Secondary Outcome: Change From Baseline Between, Gralise® and Neurontin®, Gralise® and Lyrica® for Cognitive Evaluation of Cogstate - One Card Learning (OCLT).
Description: Cogstate - The One Card Learning Test (OCLT) is a measure of visual learning and uses a well-validated pattern separation paradigm with playing card stimuli. Higher Score is better performance. Higher change from baseline means better performance.
Time Frame: Baseline and Hour 3 on Day 3
Measure: Least Squares Mean (Standard Error); unit: Score on Scale
Arm/Group | Gralise® (Gabapentin) | Neurontin® (Gabapentin) | Lyrica® (Pregabalin) | Placebo (Sugar Pill)
Number analyzed (Participants) | 28 | 31 | 30 | 30
Score on Scale | 0.02 (0.021) | 0.06 (0.020) | 0.00 (0.020) | 0.03 (0.020)
Statistical Analysis 1: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Test type: Superiority; p = 0.0070, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.08 to -0.01], Standard Error of Mean 0.0175 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 2: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Test type: Superiority; p = 0.5183, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.02 to 0.05], Standard Error of Mean 0.0175 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 3: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Test type: Superiority; p = 0.5084, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.05 to 0.02], Standard Error of Mean 0.0175 — SE of difference estimated by dividing width of 95% CI by 4

8. Secondary Outcome: Change From Baseline Between, Gralise® and Neurontin®, Gralise® and Lyrica® for Sedation Evaluation - Karolinska Sleepiness Scale (KSS).
Description: Scale: 1-9, 1=extremely alert, 9 = very sleepy, great effort to keep awake, fighting sleep
Time Frame: Baseline and Hour 3 on Day 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Gralise® (Gabapentin) | Neurontin® (Gabapentin) | Lyrica® (Pregabalin) | Placebo (Sugar Pill)
Number analyzed (Participants) | 28 | 31 | 30 | 30
units on a scale | .774 (.2985) | .264 (.2876) | .868 (.2913) | .264 (.2914)
Statistical Analysis 1: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Test type: Superiority; p = 0.1026, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.510, 95% CI 2-sided [-0.104 to 1.124], Standard Error of Mean 0.307 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 2: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Test type: Superiority; p = 0.7634, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.094, 95% CI 2-sided [-0.711 to 0.523], Standard Error of Mean 0.309 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 3: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Test type: Superiority; p = 0.1041, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.510, 95% CI 2-sided [-0.107 to 1.127], Standard Error of Mean 0.309 — SE of difference estimated by dividing width of 95% CI by 4

9. Secondary Outcome: Change From Baseline Between, Gralise® and Neurontin®, Gralise® and Lyrica® for Sedation Evaluation - Portland Neurotoxicity Scale (PNS).
Description: Portland Neurotoxicity Scale (PNS) comprises 15 questions measured on a 10-point scale. [1=No problem, 2, 3, 4, 5=Often a problem, 6, 7, 8, 9, 10=Severe problem] in 16 categories. Each question was analyzed and is presented in the same way as the primary endpoints.
Time Frame: Baseline and Hour 3 on Day 3
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Gralise® (Gabapentin) | Neurontin® (Gabapentin) | Lyrica® (Pregabalin) | Placebo (Sugar Pill)
Number analyzed (Participants) | 31 | 31 | 31 | 31
scores on a scale
  Vision (blurring, double vision): number analyzed (Participants) | 28 | 31 | 30 | 30
  Vision (blurring, double vision) | 0.036 (0.1274) | 0.322 (0.1235) | 0.249 (0.1249) | 0.115 (0.1249)
  Energy Level (get up and go): number analyzed (Participants) | 28 | 31 | 30 | 30
  Energy Level (get up and go) | 0.099 (0.1811) | 0.256 (0.1743) | 0.315 (0.1766) | 0.331 (0.1766)
  Memory (ability to remember people, places, or thi: number analyzed (Participants) | 28 | 31 | 30 | 30
  Memory (ability to remember people, places, or thi | 0.077 (0.1498) | 0.123 (0.1441) | 0.125 (0.1460) | -0.041 (0.1460)
  Walking (balance): number analyzed (Participants) | 28 | 31 | 30 | 30
  Walking (balance) | 0.206 (0.1245) | 0.327 (0.1187) | 0.405 (0.1206) | 0.107 (0.1206)
  Interest (in activities): number analyzed (Participants) | 28 | 31 | 30 | 30
  Interest (in activities) | 0.046 (0.1174) | 0.030 (0.1130) | 0.096 (0.1145) | 0.070 (0.1145)
  Coordination: number analyzed (Participants) | 28 | 31 | 30 | 30
  Coordination | 0.180 (0.1338) | 0.392 (0.1289) | 0.350 (0.1306) | 0.218 (0.1306)
  Tremor (shakiness): number analyzed (Participants) | 28 | 30 | 30 | 30
  Tremor (shakiness) | -0.103 (0.0571) | 0.037 (0.0555) | -0.031 (0.0556) | 0.068 (0.0556)
  Concentration (ability to concentrate on a task): number analyzed (Participants) | 28 | 31 | 30 | 30
  Concentration (ability to concentrate on a task) | 0.080 (0.1205) | 0.164 (0.1148) | 0.137 (0.1166) | 0.182 (0.1166)
  Speech (slurring words): number analyzed (Participants) | 28 | 31 | 30 | 30
  Speech (slurring words) | 0.035 (0.0516) | 0.133 (0.0493) | 0.065 (0.0501) | 0.103 (0.0501)
  Forgetfulness: number analyzed (Participants) | 28 | 31 | 30 | 30
  Forgetfulness | 0.118 (0.1128) | 0.227 (0.1083) | 0.175 (0.1098) | 0.079 (0.1099)
  Sleepiness (fatigue, sedation, tiredness): number analyzed (Participants) | 28 | 31 | 30 | 30
  Sleepiness (fatigue, sedation, tiredness) | 0.693 (0.2928) | 0.635 (0.2802) | 1.176 (0.2843) | 0.541 (0.2844)
  Moodiness: number analyzed (Participants) | 28 | 31 | 30 | 30
  Moodiness | 0.181 (0.1174) | 0.163 (0.1144) | 0.098 (0.1155) | 0.100 (0.1155)
  Alertness: number analyzed (Participants) | 28 | 31 | 30 | 30
  Alertness | 0.297 (0.1854) | 0.451 (0.1786) | 0.607 (0.1809) | 0.353 (0.1809)
  Attention Span: number analyzed (Participants) | 28 | 31 | 30 | 30
  Attention Span | 0.020 (0.1115) | 0.133 (0.1070) | 0.146 (0.1085) | 0.015 (0.1085)
  Motivation: number analyzed (Participants) | 28 | 31 | 30 | 30
  Motivation | 0.185 (0.1338) | 0.232 (0.1294) | 0.368 (0.1309) | 0.271 (0.1309)
Statistical Analysis 1: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Vision; Test type: Superiority; p = 0.0177, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.286, 95% CI 2-sided [-0.521 to -0.051], Standard Error of Mean 0.12 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 2: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Energy Level; Test type: Superiority; p = 0.4120, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.157, 95% CI 2-sided [-0.536 to 0.222], Standard Error of Mean 0.19 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 3: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Memory; Test type: Superiority; p = 0.7724, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.046, 95% CI 2-sided [-0.362 to 0.270], Standard Error of Mean 0.16 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 4: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Walking Balance; Test type: Superiority; p = 0.4255, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.121, 95% CI 2-sided [-0.423 to 0.180], Standard Error of Mean 0.15 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 5: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Interest in activities; Test type: Superiority; p = 0.8925, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.017, 95% CI 2-sided [-0.229 to 0.262], Standard Error of Mean 0.12 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 6: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Coordination; Test type: Superiority; p = 0.1293, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.212, 95% CI 2-sided [-0.487 to 0.063], Standard Error of Mean 0.14 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 7: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Tremor; Test type: Superiority; p = 0.0304, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.140, 95% CI 2-sided [-0.266 to -0.014], Standard Error of Mean 0.06 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 8: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Concentration; Test type: Superiority; p = 0.5811, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.084, 95% CI 2-sided [-0.384 to 0.217], Standard Error of Mean 0.15 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 9: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Speech; Test type: Superiority; p = 0.1144, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.098, 95% CI 2-sided [-0.220 to 0.024], Standard Error of Mean 0.06 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 10: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Forgetfulness; Test type: Superiority; p = 0.3774, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.109, 95% CI 2-sided [-0.352 to 0.135], Standard Error of Mean 0.12 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 11: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Sleepiness; Test type: Superiority; p = 0.8658, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.057, 95% CI 2-sided [-0.613 to 0.727], Standard Error of Mean 0.34 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 12: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Moodiness; Test type: Superiority; p = 0.8543, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.018, 95% CI 2-sided [-0.179 to 0.216], Standard Error of Mean 0.10 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 13: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Alertness; Test type: Superiority; p = 0.4294, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.153, 95% CI 2-sided [-0.537 to 0.231], Standard Error of Mean 0.19 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 14: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Attention Span; Test type: Superiority; p = 0.3613, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.113, 95% CI 2-sided [-0.357 to 0.132], Standard Error of Mean 0.12 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 15: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Motivation; Test type: Superiority; p = 0.7201, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.047, 95% CI 2-sided [-0.305 to 0.212], Standard Error of Mean 0.13 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 16: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Vision; Test type: Superiority; p = 0.0767, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.213, 95% CI 2-sided [-0.448 to 0.023], Standard Error of Mean 0.12 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 17: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Energy Level; Test type: Superiority; p = 0.2618, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.216, 95% CI 2-sided [-0.597 to 0.165], Standard Error of Mean 0.19 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 18: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Memory; Test type: Superiority; p = 0.7633, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.048, 95% CI 2-sided [-0.366 to 0.269], Standard Error of Mean 0.16 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 19: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Walking Balance; Test type: Superiority; p = 0.1968, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.198, 95% CI 2-sided [-0.502 to 0.105], Standard Error of Mean 0.15 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 20: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Interest in Activities; Test type: Superiority; p = 0.6891, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.050, 95% CI 2-sided [-0.296 to 0.197], Standard Error of Mean 0.12 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 21: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Coordination; Test type: Superiority; p = 0.2229, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.171, 95% CI 2-sided [-0.447 to 0.106], Standard Error of Mean 0.14 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 22: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Tremor; Test type: Superiority; p = 0.2591, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.072, 95% CI 2-sided [-0.197 to 0.054], Standard Error of Mean 0.06 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 23: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Concentration; Test type: Superiority; p = 0.7099, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.057, 95% CI 2-sided [-0.359 to 0.246], Standard Error of Mean 0.15 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 24: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Speech; Test type: Superiority; p = 0.6215, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.031, 95% CI 2-sided [-0.154 to 0.092], Standard Error of Mean 0.06 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 25: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Forgetfulness; Test type: Superiority; p = 0.6422, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.057, 95% CI 2-sided [-0.302 to 0.187], Standard Error of Mean 0.12 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 26: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Sleepiness; Test type: Superiority; p = 0.1574, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.483, 95% CI 2-sided [-1.157 to 0.190], Standard Error of Mean 0.34 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 27: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Moodiness; Test type: Superiority; p = 0.4039, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.084, 95% CI 2-sided [-0.115 to 0.282], Standard Error of Mean 0.10 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 28: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Alertness; Test type: Superiority; p = 0.1145, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.309, 95% CI 2-sided [-0.695 to 0.076], Standard Error of Mean 0.19 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 29: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Attention Span; Test type: Superiority; p = 0.3083, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.127, 95% CI 2-sided [-0.372 to 0.119], Standard Error of Mean 0.12 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 30: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Motivation; Test type: Superiority; p = 0.1638, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.183, 95% CI 2-sided [-0.443 to 0.0776], Standard Error of Mean 0.13 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 31: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Vision; Test type: Superiority; p = 0.5101, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.078, 95% CI 2-sided [-0.314 to 0.157], Standard Error of Mean 0.12 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 32: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Energy Level; Test type: Superiority; p = 0.2285, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.233, 95% CI 2-sided [-0.614 to 0.149], Standard Error of Mean 0.19 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 33: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Memory; Test type: Superiority; p = 0.4612, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.118, 95% CI 2-sided [-0.200 to 0.436], Standard Error of Mean 0.16 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 34: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Walking Balance; Test type: Superiority; p = 0.5190, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.099, 95% CI 2-sided [-0.205 to 0.402], Standard Error of Mean 0.15 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 35: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Interest in Activities; Test type: Superiority; p = 0.8479, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.024, 95% CI 2-sided [-0.271 to 0.223], Standard Error of Mean 0.12 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 36: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Coordination; Test type: Superiority; p = 0.7808, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.039, 95% CI 2-sided [-0.316 to 0.238], Standard Error of Mean 0.14 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 37: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Tremor; Test type: Superiority; p = 0.0083, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.171, 95% CI 2-sided [-0.296 to -0.045], Standard Error of Mean 0.06 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 38: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Concentration; Test type: Superiority; p = 0.5068, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.101, 95% CI 2-sided [-0.404 to 0.201], Standard Error of Mean 0.15 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 39: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Speech; Test type: Superiority; p = 0.2725, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.068, 95% CI 2-sided [-0.191 to 0.055], Standard Error of Mean 0.06 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 40: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Forgetfulness; Test type: Superiority; p = 0.7498, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.039, 95% CI 2-sided [-0.206 to 0.284], Standard Error of Mean 0.12 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 41: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Sleepiness; Test type: Superiority; p = 0.6554, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.152, 95% CI 2-sided [-0.522 to 0.826], Standard Error of Mean 0.34 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 42: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Moodiness; Test type: Superiority; p = 0.4143, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.082, 95% CI 2-sided [-0.116 to 0.280], Standard Error of Mean 0.10 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 43: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Alertness; Test type: Superiority; p = 0.7761, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.055, 95% CI 2-sided [-0.441 to 0.330], Standard Error of Mean 0.19 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 44: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Attention Span; Test type: Superiority; p = 0.9697, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.005, 95% CI 2-sided [-0.241 to 0.251], Standard Error of Mean 0.12 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 45: Comparison: Gralise® (Gabapentin) vs Placebo (Sugar Pill); Motivation; Test type: Superiority; p = 0.5118, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.086, 95% CI 2-sided [-0.346 to 0.174], Standard Error of Mean 0.13; SE of difference estimated by dividing width of 95% CI by 4

10. Secondary Outcome: Change From Baseline Between Gralise® and Neurontin® in the Driving Simulator - Standard Deviation of Vehicle Speed (SDVS).
Description: Miles per Hour (mph)
Time Frame: Baseline and Hour 3 on Day 3
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mph
Arm/Group | Gralise® (Gabapentin) | Neurontin® (Gabapentin) | Placebo
Number analyzed (Participants) | 28 | 31 | 30
mph | 0.831 (0.4844) | 0.947 (0.4648) | 0.851 (0.4715)
Statistical Analysis 1: Comparison: Gralise® (Gabapentin) vs Neurontin® (Gabapentin); Test type: Superiority; p = 0.8293, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.116, 95% CI 2-sided [-1.178 to 0.947], Standard Error of Mean 0.53 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 2: Comparison: Gralise® (Gabapentin) vs Placebo; Test type: Superiority; p = 0.9705, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.020, 95% CI 2-sided [-1.089 to 1.049], Standard Error of Mean 0.53 — SE of difference estimated by dividing width of 95% CI by 4

11. Secondary Outcome: Change From Baseline Between Gralise® and Lyrica® in the Driving Simulator - Standard Deviation of Vehicle Speed (SDVS).
Description: Miles per Hour (mph)
Time Frame: Baseline and Hour 3 on Day 3
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mph
Arm/Group | Gralise® (Gabapentin) | Lyrica® (Pregabalin) | Placebo
Number analyzed (Participants) | 28 | 30 | 30
mph | 0.831 (0.4844) | 1.319 (0.4713) | 0.851 (0.4715)
Statistical Analysis 1: Comparison: Gralise® (Gabapentin) vs Lyrica® (Pregabalin); Test type: Superiority; p = 0.3666, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.488, 95% CI 2-sided [-1.556 to 0.581], Standard Error of Mean 0.53 — SE of difference estimated by dividing width of 95% CI by 4
Statistical Analysis 2: Comparison: Gralise® (Gabapentin) vs Placebo; Test type: Superiority; p = 0.9705, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.020, 95% CI 2-sided [-1.089 to 1.049], Standard Error of Mean 0.53 — SE of difference estimated by dividing width of 95% CI by 4

12. Secondary Outcome: To Compare the Relative Safety and Tolerability of Gralise®, Neurontin®, and Lyrica®.
Description: * Number of subjects with Treatment-Emergent Adverse Events (TEAE)
  * Number of subjects with Serious Adverse Event (SAE)
  * Number of subjects discontinued due to Adverse Event (AE)
Time Frame: Screening to 1 week after Period 4 discharge
Measure: Number; unit: participants
Groups:
- Placebo (Sugar Pill): Placebo (sugar pill): Three (3) placebo tablets matching the appearance of Gralise® & 1 placebo capsule matching the over-encapsulation of doses of Neurontin® & Lyrica®.
Arm/Group | Gralise® (Gabapentin) | Neurontin® (Gabapentin) | Lyrica® (Pregabalin) | Placebo (Sugar Pill)
Number analyzed (Participants) | 28 | 31 | 31 | 30
participants
  Subjects with TEAE | 6 | 13 | 16 | 5
  Subjects with SAE | 0 | 0 | 0 | 0
  Subjects Discontinued due to AE | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: 7 weeks
Description: Adverse Events were reported from the signed informed consent to 30 days after the last dose of study drug.
Arm/Group | Gralise® (Gabapentin) | Neurontin® (Gabapentin) | Lyrica® (Pregabalin) | Placebo (Sugar Pill)
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/31 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 6/28 | 11/31 | 14/31 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gralise® (Gabapentin) (N=28) | Neurontin® (Gabapentin) (N=31) | Lyrica® (Pregabalin) (N=31) | Placebo (Sugar Pill) (N=30)
Somnolence (Nervous system disorders) | 3 | 7 | 4 | 1
Dizziness (Nervous system disorders) | 3 | 4 | 6 | 0
Headache (Nervous system disorders) | 1 | 0 | 5 | 1
Euphoric mood (Psychiatric disorders) | 1 | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees that sponsor shall have the right to the first publication of the study results which is intended to be a joint, multi-center publication. Following the first publication, the PI may publish study data or results, provided however PI submits the proposed publication to sponsor for review at least 60 days prior to the date of the proposed publication. Sponsor may remove any information that is considered confidential and / or proprietary other than study data.